CLINICAL TRIAL: NCT05659979
Title: The Role of Comprehensive Geriatric Assessment in Older Patients Affected by Knee Osteoarthritis: an Exploratory Randomized Controlled Trial
Brief Title: Comprehensive Geriatric Assessment in Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Palermo (Other)
Collaborators: Charles University, Czech Republic (Other); Ente Ospedaliero Ospedali Galliera (Other); St. Marien-Hospital Düren (Other); Erasmus University Rotterdam (Other)
Responsible Party: Principal Investigator, Nicola Veronese, Dr., University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITA7976
Record Dates: First submitted 2022-12-03; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Osteo Arthritis Knee
MeSH Terms: interventions — Geriatric Assessment

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Geriatric Assessment (Experimental): This group will receive a comprehensive geriatric assessment evaluation during the study, using the multidimensional prognostic index
  Interventions: Other: Comprehensive geriatric assessment
- Controls (No Intervention): This group will receive standard/usual care

INTERVENTIONS:
Other: Comprehensive geriatric assessment — A detailed comprehensive geriatric assessment will be given to all the participants randomized to this group, including the administration of multidimensional prognostic index (MPI), a tool derived from the CGA and consisting of eight different domains.
  Arms: Comprehensive Geriatric Assessment

SUMMARY:
Osteoarthritis (OA) is the most common form of arthritis, and is characterized by joint pain and stiffness leading to functional decline and relevant loss in quality of life. The management of knee OA is demanded to several specialists, including general practitioners, rheumatologists, orthopedics and finally geriatricians. However, the exact role of geriatricians in the management of knee OA was poorly studied, whilst the comprehensive geriatric assessment (CGA) is widely used for preventing negative consequences in older people.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common form of arthritis, and is characterized by joint pain and stiffness leading to functional decline and relevant loss in quality of life. The incidence of OA is rising due to the aging population and an increase in some risk factors, such as obesity. Knee OA is the most common OA localization, and symptomatic knee OA is highly prevalent among people aged over 50 years, affecting more than 250 million people worldwide.

Knee OA is a leading cause of pain in older people, and pain of the hip and knee results in physical disability and an increased risk of all-cause mortality. Hip and knee OA together are the eleventh highest contributor to global disability: the years of life lived with OA-related disability increased by 64% from 1990 to 2010 reaching 17 million. OA is a progressive disorder, with different degrees of severity, that requires long-term management with various treatment options over the course of the disease. The goals of treatment for OA are to reduce symptoms and ultimately slow disease progression, which may in turn reduce the impact of OA on the patient's mobility and quality of life, with consequent reduction in healthcare resource needs.

In 2019, the European Society for Clinical and Economic Aspects of Osteoporosis, Osteoarthritis and Musculoskeletal Diseases (ESCEO) published recommendations for the management of knee OA in the form of a treatment algorithm that provides practical guidance for the prioritization of interventions and guides physicians through progressive, logical steps based on the severity of the knee OA signs/symptoms.

The management of knee OA is therefore demanded to several specialists, including general practitioners, rheumatologists, orthopedics and finally geriatricians. However, the exact role of geriatricians in the management of knee OA was poorly studied, whilst the comprehensive geriatric assessment (CGA) is widely used for preventing negative consequences in older people, such as hospitalization or mortality. Moreover, CGA can be used across different settings, from primary care to hospital, with similar beneficial effects in older people. Finally, people affected by knee OA are usually affected by other medical (e.g., dementia, cardiovascular diseases, depression) and non-medical (e.g., loneliness) conditions that can limit the adherence to therapeutic approaches, therefore limiting the efficacy of the interventions suggested in knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age > 70 years; able to sign the informed consent
* Diagnosis of knee OA according to standardized criteria in Grade 1 (doubtful narrowing of joint space and possible osteophytic lipping), Grade 2 (definite osteophytes and possible narrowing of joint space) Kellgren and Lawrence system or Grade 3 (moderate multiple osteophytes, definite narrowing of joint space and some sclerosis and possible deformity of bone ends).

Exclusion Criteria:

* Expected life expectancy less than 6 months
* Previous orthopedic surgery, in the three months before the enrolment or a planned orthopedic intervention in the next 6 months.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain, physical function, stiffness | Baseline, 3 months, 6 months
  We will use the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scale. The WOMAC, that is one of the most used tool in knee OA research, measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). The single items of the WOMAC will be assessed as co-primary outcomes.

SECONDARY OUTCOMES:
Change in the adherence to medications | Baseline, 3 months, 6 months
  Adherence to medications suggested during the first visit will be evaluated during the follow-up period using questionnaires.
Change in the severity of multidimensional frailty | Baseline, 3 months, 6 months
  This outcome will be explored using the multidimensional prognostic index (MPI), a scale that measures eight different domains typical of older people. The sum of the calculated scores from the eight domains will be divided by 8 to obtain a final MPI risk score ranging from 0 = no risk to 1 = higher risk of mortality.
Change in the quality of life | Baseline, 3 months, 6 months
  The short form 36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the less quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Veronese, MD, Principal Investigator — University of Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Veronese N, Fazzari A, Santangelo E, Iommi C, Soysal P, Custodero C, Pickert L, Polidori MC, Stolniceanu N, Michalkova H, Topinkova E, Pilotto A, Barbagallo M. The role of comprehensive geriatric assessment in older patients affected by knee osteoarthritis: an exploratory randomized controlled trial. Aging Clin Exp Res. 2025 May 16;37(1):155. doi: 10.1007/s40520-025-03061-0. PMID 40377819